CLINICAL TRIAL: NCT04517084
Title: A Retroactive Study on the Motivations of Patients Undergoing Bariatric Surgery
Brief Title: Pre-surgical Motivation for Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: YNC2MCIRS
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2018-10

CONDITIONS: Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study investigating the motivations of patients who had undergone bariatric surgery using data collected from questionnaires given to patients prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergone bariatric surgery at Singapore General Hospital and completed the life center questionnaire.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Undergone bariatric surgery within SGH LIFE Centre and completed the intake questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 5 years post surgery
  Weight Loss in Kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore